CLINICAL TRIAL: NCT02637973
Title: Effects of Empagliflozin on Liver Fat Content, Energy Metabolism and Body Composition in Patients With Type 2 Diabetes
Acronym: EmLiFa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Deutsche Diabetes Forschungsgesellschaft e.V. (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Organization: German Diabetes Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EmLiFa001
Record Dates: First submitted 2015-12-16; First posted 2015-12-22 (Estimated); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Type 2 Diabetes; Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Empagliflozin (Experimental): Empagliflozin, film-tablet, 25mg once daily
  Interventions: Drug: Empagliflozin
- Placebo (Placebo Comparator): Placebo, once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin — 25 mg once daily
  Other Names: Jardiance
  Arms: Empagliflozin
Drug: Placebo — once daily
  Other Names: No Drug Therapy
  Arms: Placebo

SUMMARY:
The effects of empagliflozin treatment on hepatocellular lipid content, liver energy metabolism and body composition will be investigated in a multicentre, prospective, placebo-controlled, double-blind, randomized, 2-arm parallel, interventional and exploratory pilot study in patients with newly diagnosed type 2 diabetes.

DETAILED DESCRIPTION:
In this multicentre, prospective, placebo-controlled, double-blind, randomized, 2-arm parallel, interventional pilot study HCL and intramyocellular lipids (IMCL) will be quantified with 1H magnetic resonance (MR) spectroscopy. Hepatic ATP and inorganic phosphate (Pi) concentrations will be assessed with 31P MR spectroscopy (1). Whole-body and hepatic insulin sensitivity and metabolic flexibility will be measured by combining hyperinsulinemic-euglycemic pancreatic clamp tests with isotopic dilution of 6,6-2H2 glucose and indirect calorimetry as shown (2). Abdominal fat distribution will be quantified by MR imaging.

Newly diagnosed patients with type 2 diabetes (T2D) will be randomly allocated to once daily 25 mg empagliflozin (EMPA) or placebo for 24 weeks with a computer-generated random sequence and will be masked to the treatment assignment. Participants will visit the clinical research center at baseline, 12 weeks and 24 weeks for MRS and metabolic examinations, including blood sampling for hepato- and adipocytokines. Anthropometric parameters (body weight, waist circumference, total body fat, blood pressure) and glycemic control (HbA1C, fasting blood glucose, FBG) will be assessed at baseline and during monitoring visits every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years
* BMI<45 kg/m2
* known diabetes duration up to 7 years
* 6%≤HbA1c≤8%
* drug naïve - no previous antihyperglycemic treatment or one month washout period of treatment with oral glucose lowering drugs (no previous treatment with thiazolidinedione (TZD) drugs allowed)
* obtained written informed consent

Exclusion Criteria:

* uncontrolled hyperglycaemia at screening (glucose level ≥240 mg/dl after an overnight fast, confirmed by a second measurement)
* acute coronary syndrome, stroke or transient ischemic attack within 3 months prior to consent
* previous lower limb amputation
* severe lower limb infection/ulceration within 3 months prior to consent
* liver disease including chronic viral hepatitis (B or C), alcohol abuse, hemochromatosis, alpha-1 antitrypsin deficiency, autoimmune hepatitis, Wilson's disease, primary sclerosing cholangitis or primary biliary cirrhosis, or liver cirrhosis of any etiology
* AST or ALT > 3 x ULN
* positive result on hepatitis B (HBs-AG), hepatitis C (HCV-AB), or HIV 1 and 2 test
* impaired kidney function (estimated glomerular filtration rate [eGFR]<60 mL/min/1.73m2) during screening
* structural and functional urogenital abnormalities, that predispose for urogenital infections
* gastrointestinal surgeries that induce chronic malabsorption
* history of cancer (except basal cell carcinoma) or treatment for cancer within 5 years
* blood dyscrasias or any disorders causing haemolysis or unstable erythrocytes
* treatment with antiobesity drugs 3 months prior to consent
* treatment with immunomodulatory drugs (oral steroids, antihistamines)
* change in dosage of thyroid hormones within 6 weeks of consent
* pregnancy, lactation period
* metal or magnetic implants, devices or objects inside of or on the body, which are not MRI compatible (according to MRT safety checklist in Appendix 11.3)
* claustrophobia
* cigarette smoking (non-smoker < 1year), alcohol consumption (male >30 g/d, female >20g/d)
* drug abuse or psychiatric disease
* night-worker or circumstances not allowing normal day-night rhythm
* hypersensitivity to empagliflozin (or drugs of similar chemical structure) or any of the drug compounds
* pharmaceutical preparations with which interactions can be expected - amiloride, furosemide, indapamide, spironolactone, torasemide, triamterene
* use of anti-NASH drugs (vitamin E, ursodeoxycholic acid, S-adenosylmethionine, betaine, silymarin, gemfibrozil, anti-TNF therapies, probiotics) in the 3 months prior to randomization
* women of childbearing potential not using two adequate methods of contraception including a barrier method and a highly efficacious non-barrier method
* persons with any kind of dependency on the investigator or employed by the sponsor or investigator
* persons held in an institution by legal or official order
* participation in another trial in the last 10 weeks before randomization or planned participation during the trial period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-12; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Change in liver fat content | from baseline to 24 weeks
  Change in liver fat content between baseline and 24 weeks measured with magnetic resonance spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, MD, Principal Investigator — Deutsches Diabetes Zentrum
Locations (5):
- Germany (5):
  - Charite Universitaetsmedizin Berlin, Berlin
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden
  - German Diabetes Center, Düsseldorf
  - University Clinic Heidelberg, Heidelberg
  - University Clinic Tübingen, Tübingen